CLINICAL TRIAL: NCT00535847
Title: A Phase 2 Rollover Protocol of Telaprevir (VX-950) in Combination With Peginterferon Alfa-2a (Pegasys®) and Ribavirin (Copegus®) in Subjects Enrolled in the Control Group (Group A) of Study VX06-950-106, VX05-950-104 and VX05-950-104EU Who Did Not Achieve or Maintain an Undetectable HCV RNA Level Through Sustained Viral Response
Brief Title: A Rollover Study for Subjects Participating in the Control Arm of Study VX06-950-106, VX05-950-104 and VX05-950-104EU Whose Plasma Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) Levels Did Not Respond to Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Collaborators: Tibotec, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VX06-950-107
Record Dates: First submitted 2007-09-25; First posted 2007-09-26 (Estimated); Results first posted 2011-07-25 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-07

CONDITIONS: Hepatitis C
Keywords: Genotype 1
MeSH Terms: conditions — Hepatitis C | interventions — telaprevir; Ribavirin; peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 24 Week (Experimental): Telaprevir 750 mg tablet thrice daily for 12 weeks in combination with pegylated interferon alfa 2a (Peg-IFN-alfa-2a) 180 microgram per week (mcg/week) subcutaneous injection and ribavirin (RBV) tablet orally twice daily at a dose of 1000 milligram per day (mg/day) for subjects weighing less than (<) 75 kilogram (kg) and 1200 mg/day for subjects weighing greater than or equal to (>=) 75 kg, for 24 weeks.
  Interventions: Drug: Telaprevir; Drug: Ribavirin; Drug: Pegylated interferon alfa 2a
- Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 48 Week (Experimental): Telaprevir 750 mg tablet thrice daily for 12 weeks in combination with Peg-IFN-alfa-2a 180 mcg/week subcutaneous injection and RBV tablet orally twice daily at a dose of 1000 mg/day for subjects weighing <75 kg and 1200 mg/day for subjects weighing >=75 kg, for 48 weeks.
  Interventions: Drug: Telaprevir; Drug: Ribavirin; Drug: Pegylated interferon alfa 2a
- Other (Experimental): Subjects received telaprevir 750 mg tablet thrice daily in combination with Peg-IFN-alfa-2a 180 mcg/week subcutaneous injection and RBV tablet orally twice daily at a dose of 1000 mg/day for subjects <75 kg and 1200 mg/day for subjects weighing >=75 kg, discontinued treatment before Week 12 in this study (VX06-950-107 [NCT00535847]) and had a partial response, viral breakthrough, or relapse in the parent study (VX05-950-104 [NCT00336479], VX05-950-104EU [NCT00372385] or VX06-950-106 [NCT00420784]) were included in "Other" reporting group.
  Interventions: Drug: Telaprevir; Drug: Ribavirin; Drug: Pegylated interferon alfa 2a

INTERVENTIONS:
Drug: Telaprevir — Tablet
  Other Names: VX-950
Drug: Ribavirin — Tablet
Drug: Pegylated interferon alfa 2a — Solution for Injection

SUMMARY:
To provide access to a telaprevir-based treatment to subjects of the Control Group of Study VX06-950-106 (NCT00420784), VX05-950-104 (NCT00336479), and VX05-950-104EU (NCT00372385) who stopped treatment due to inadequate response to treatment. Safety, tolerability, and Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) levels will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the control arm of Study VX06-950-106 (NCT00420784), VX05-950-104 (NCT00336479) or VX05-950-104EU (NCT00372385)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2007-10; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Adda, MD, Study Director — Vertex Pharmaceuticals Incorporated
Locations (62):
- United States (39):
  - Birmingham, Alabama
  - Los Angeles, California
  - Kaiser Permanente Internal Medicine, San Diego, California
  - San Francisco, California
  - University of Colorado Health Sciences Center, Denver, Colorado
  - South Denver Gastroenterology, Englewood, Colorado
  - University of Florida, Gainesville, Florida
  - Borland-Groover Clinic, Jacksonville, Florida
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - University of Miami Center for Liver Diseases, Miami, Florida
  - Sarasota, Florida
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Indianapolis, Indiana
  - Digestive and Liver Disease Clinic, Baton Rouge, Louisiana
  - Virology Treatment Center, Maine Medical Center, Portland, Maine
  - Johns Hopkins University, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - St Louis University, St Louis, Missouri
  - The Nebraska Medical Center, Omaha, Nebraska
  - University of New Mexico, Albuquerque, New Mexico
  - North Shore University Hospital, Manhasset, New York
  - New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland, Ohio
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Columbia Gastroenterology Associates, PA, Columbia, South Carolina
  - Memphis Gastroenterology Group, Germantown, Tennessee
  - Liver Institute at Methodist Dallas, Dallas, Texas
  - Houston, Texas
  - Alamo Medical Research, San Antonio, Texas
  - Annandale, Virginia
  - University of Virginia Health Systems, Charlottesville, Virginia
  - Metropolitan Research, Fairfax, Virginia
  - McGuire DVAMC, Richmond, Virginia
- Vienna, Austria
- Canada (5):
  - University of Calgary Medical Clinic, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - University of British Columbia Vancouver General Hospital, Vancouver, British Columbia
  - Winnipeg, Manitoba
  - Toronto, Ontario
- France (6):
  - Hospital Henri Mondor, Créteil
  - Lyon
  - Nice
  - Paris
  - Pessac
  - Vandœuvre-lès-Nancy
- Germany (6):
  - Berlin
  - Universitatsklinikum Bonn, Bonn
  - University of Cologne, Cologne
  - Uniklinik Duesseldorf, Düsseldorf
  - Frankfurt
  - Hanover
- Netherlands (3):
  - Academic Medical Center, Amsterdam
  - Leiden University Medical Center, Leiden
  - Erasmus MC Medical Center, Rotterdam
- Fundacion de Investigation de Diego, Santurce, Puerto Rico
- London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects randomized to placebo control group in parent studies VX05-950-104 (NCT00336479), VX05-950-104EU (NCT00372385) and VX06-950-106 (NCT00420784) who had discontinued treatment in the parent study due to an inadequate response to treatment or relapsed after treatment were eligible to participate in this study VX06-950-107 (NCT00535847).
Period: Overall Study
Arm/Group | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 24 Week | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 48 Week | Other
Started | 81 | 34 | 2
Completed | 59 | 20 | 0
Not Completed | 22 | 14 | 2
Not completed — Adverse Event | 5 | 3 | 2
Not completed — Non compliance | 1 | 1 | 0
Not completed — Protocol-defined Virologic Stopping Rule | 16 | 10 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis (FA) set included all enrolled subjects who received at least 1 dose of study drug in this study (VX06-950-107 [NCT00535847]).
Groups:
- Total: Total of all reporting groups
Arm/Group | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 24 Week | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 48 Week | Other | Total
Number analyzed (Participants) | 81 | 34 | 2 | 117
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 81 | 34 | 2 | 117
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.0 (7.7) | 51.2 (5.9) | 49.0 (0.0) | 50.3 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 8 | 0 | 36
  Male | 53 | 26 | 2 | 81
Region of Enrollment [Number; unit: participants]
  North America | 64 | 26 | 2 | 92
  Europe | 17 | 8 | 0 | 25

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Undetectable Plasma Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) at Week 24 After the Completion of Treatment
Description: The plasma HCV RNA level was measured using Roche TaqMan HCV RNA assay. The lower limit of detection was 10 international units per milliliter (IU/mL).
Time Frame: 24 weeks after the completion of treatment (up to Week 72)
Population: The FA set included all enrolled subjects who received at least 1 dose of study drug in this study (VX06-950-107 [NCT00535847]).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 24 Week | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 48 Week | Other
Number analyzed (Participants) | 81 | 34 | 2
percentage of participants | 60.5 [49.0 to 71.2] | 52.9 [35.1 to 70.2] | 100.0 [15.8 to 100.0]

2. Secondary Outcome: Percentage of Prior Relapsers With Undetectable HCV RNA
Description: Prior relapsers: subjects who had undetectable HCV RNA at the end of treatment in parent study but reverted to detectable levels of HCV RNA after stopping treatment in parent study were categorized as prior relapsers. Percentage of prior relapsers with undetectable HCV RNA 24 weeks after the completion of treatment in this study were presented. The plasma HCV RNA level was measured using Roche TaqMan HCV RNA assay. The lower limit of detection was 10 international units per milliliter (IU/mL).
Time Frame: 24 weeks after the completion of treatment (up to Week 72)
Population: Analysis population included all enrolled subjects who were prior relapsers in parent study (VX05-950-104 [NCT00336479], VX05-950-104EU [NCT00372385] or VX06-950-106 [NCT00420784]) and received at least 1 dose of study drug in this study (VX06-950-107 [NCT00535847]).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 24 Week | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 48 Week | Other
Number analyzed (Participants) | 25 | 3 | 1
percentage of participants | 96.0 [79.6 to 99.9] | 100.0 [29.2 to 100.0] | 100.0 [2.5 to 100.0]

3. Secondary Outcome: Percentage of Subjects With End of Treatment Response
Description: Subjects were considered to have an end of treatment response if they completed the assigned treatment regimen and had undetectable HCV RNA at end of treatment or prematurely discontinued the assigned treatment regimen and had undetectable HCV RNA at the time of discontinuation. The plasma HCV RNA level was measured using Roche TaqMan HCV RNA assay. The lower limit of detection was 10 international units per milliliter (IU/mL).
Time Frame: End of treatment (up to Week 48)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 24 Week | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 48 Week | Other
Number analyzed (Participants) | 81 | 34 | 2
percentage of participants | 72.8 [61.8 to 82.1] | 64.7 [46.5 to 80.3] | 100.0 [15.8 to 100.0]

4. Secondary Outcome: Percentage of Subjects With Undetectable HCV RNA at Week 48 After Completion of Treatment Among Subjects Who Completed Assigned Treatment
Description: as for outcome 1
Time Frame: 48 weeks after completion of treatment (up to Week 96)
Population: Analysis population included subjects who completed assigned treatment in this study (VX06-950-107 [NCT00535847]).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 24 Week | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 48 Week | Other
Number analyzed (Participants) | 59 | 20 | 0
percentage of participants | 83.1 [71.0 to 91.6] | 70.0 [45.7 to 88.1] |

5. Secondary Outcome: Cross Tabulation of Extended Rapid Viral Response (eRVR) and Sustained Viral Response (SVR) in With Prior Response
Description: Cross tabulation of number of subjects with eRVR/SVR status in present study was presented with respect to prior response status of subjects in parent studies. eRVR=undetectable HCV RNA at Week 4 and Week 12, SVR=undetectable HCV RNA at end of treatment (EOT) and at 24 weeks after last dose of study treatment without any confirmed detectable HCV RNA in between. Prior response=subjects were categorized into following categories based on their viral response in the parent study: Null Response (less than [<] 1-log10 decrease in HCV RNA at Week 4 or <2-log10 decrease in HCV RNA at Week 12), Partial Response (greater than [>] 2-log10 decrease in HCV RNA at Week 12, but detectable HCV RNA at Week 24), Viral Breakthrough (detectable HCV RNA during treatment after achieving undetectable HCV RNA), Relapse (undetectable HCV RNA at EOT but detectable HCV RNA during viral follow-up). Plasma HCV RNA level was measured using Roche TaqMan HCV RNA assay; lower limit of detection=10 IU/mL.
Time Frame: Baseline up to Week 72
Population: The FA set included subjects who received at least 1 dose of study drug in this study (VX06-950-107 [NCT00535847]). Data was presented for overall subjects based on eRVR and SVR status as per planned analysis.
Measure: Number; unit: participants
Groups:
- Achieved eRVR/Achieved SVR: All subjects in "Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 24 Week", "Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 48 Week" and "Other" reporting groups who achieved eRVR and SVR in this study (VX06-950-107 [NCT00535847]).
- Achieved eRVR/Did Not Achieve SVR: All subjects in "Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 24 Week", "Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 48 Week" and "Other" reporting groups who achieved eRVR but did not achieve SVR in this study (VX06-950-107 [NCT00535847]).
- Did Not Achieve eRVR/Achieved SVR: All subjects in "Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 24 Week", "Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 48 Week" and "Other" reporting groups who did not achieve eRVR but achieved SVR in this study (VX06-950-107 [NCT00535847]).
- Did Not Achieve eRVR/Did Not Achieve SVR: All subjects in "Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 24 Week", "Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 48 Week" and "Other" reporting groups who neither achieved eRVR nor SVR in this study (VX06-950-107 [NCT00535847]).
Arm/Group | Achieved eRVR/Achieved SVR | Achieved eRVR/Did Not Achieve SVR | Did Not Achieve eRVR/Achieved SVR | Did Not Achieve eRVR/Did Not Achieve SVR
Number analyzed (Participants) | 57 | 12 | 12 | 36
participants
  Prior Null Response | 12 | 5 | 7 | 27
  Prior Partial Response | 15 | 7 | 1 | 6
  Prior Viral Breakthrough | 6 | 0 | 0 | 2
  Prior Relapse | 24 | 0 | 4 | 1
Statistical Analysis 1: Comparison: Achieved eRVR/Achieved SVR vs Achieved eRVR/Did Not Achieve SVR vs Did Not Achieve eRVR/Achieved SVR vs Did Not Achieve eRVR/Did Not Achieve SVR; Stratified Analysis (Mantel-Haenszel)- The Mantel-Haenszel estimator provides an estimate of the common odds ratio for the association between eRVR and SVR across the prior response strata; Test type: Superiority or Other; Odds Ratio (OR) = 12.703, 95% CI 2-sided [4.259 to 37.884]

6. Primary Outcome: Number of Subjects With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AE: any adverse change from the subject's baseline (pre-treatment) condition, including any adverse experience, abnormal recording or clinical laboratory assessment value which occurs during the course of the study, whether it is considered related to the study drug or not. An adverse event includes any newly occurring event or previous condition that has increased in severity or frequency since the administration of study drug. SAE: medical event or condition, which falls into any of the following categories, regardless of its relationship to the study drug: death, life threatening adverse experience, in-patient hospitalization/prolongation of hospitalization, persistent/significant disability or incapacity, congenital anomaly/birth defect, important medical event. "Study drug" includes all investigational agents (including placebo, if applicable) administered during the course of the study.
Time Frame: Baseline through Week 48
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 24 Week | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 48 Week | Other
Number analyzed (Participants) | 81 | 34 | 2
participants
  AEs | 77 | 31 | 2
  SAEs | 7 | 3 | 1

ADVERSE EVENTS:
Time Frame: Adverse Events during Overall Treatment Phase (Baseline through Week 48)
Description: In the event a single participant has experienced both a serious and a non-serious form of the same adverse event term, the individual has been included in the numerator ("number of affected participants") of both adverse event tables.
Arm/Group | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 24 Week | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 48 Week | Other
Serious Adverse Events (participants affected / at risk) | 7/81 | 3/34 | 1/2
Other Adverse Events (participants affected / at risk) | 77/81 | 31/34 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 24 Week (N=81) | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 48 Week (N=34) | Other (N=2)
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Drug rash with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 3 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Bursitis infective (Infections and infestations) | 1 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 24 Week (N=81) | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 48 Week (N=34) | Other (N=2)
Fatigue (General disorders) | 30 | 21 | 1
Influenza like illness (General disorders) | 17 | 10 | 1
Pyrexia (General disorders) | 16 | 6 | 0
Chills (General disorders) | 11 | 4 | 0
Asthenia (General disorders) | 9 | 3 | 0
Injection site erythema (General disorders) | 9 | 2 | 0
Irritability (General disorders) | 6 | 4 | 1
Pain (General disorders) | 5 | 4 | 0
Oedema peripheral (General disorders) | 4 | 3 | 0
Nausea (Gastrointestinal disorders) | 20 | 11 | 1
Diarrhoea (Gastrointestinal disorders) | 19 | 6 | 0
Haemorrhoids (Gastrointestinal disorders) | 9 | 4 | 0
Anorectal discomfort (Gastrointestinal disorders) | 7 | 3 | 0
Constipation (Gastrointestinal disorders) | 3 | 6 | 0
Vomiting (Gastrointestinal disorders) | 5 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 5 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 4 | 2 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 4 | 0
Flatulence (Gastrointestinal disorders) | 0 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 34 | 9 | 2
Rash (Skin and subcutaneous tissue disorders) | 23 | 13 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 10 | 5 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 8 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 3 | 3 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 4 | 2 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 3 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Headache (Nervous system disorders) | 23 | 14 | 0
Dizziness (Nervous system disorders) | 6 | 5 | 0
Disturbance in attention (Nervous system disorders) | 2 | 2 | 0
Insomnia (Psychiatric disorders) | 14 | 7 | 1
Depression (Psychiatric disorders) | 9 | 4 | 0
Depressed mood (Psychiatric disorders) | 1 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 10 | 5 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Sinusitis (Infections and infestations) | 4 | 4 | 0
Nasopharyngitis (Infections and infestations) | 3 | 2 | 0
Urinary tract infection (Infections and infestations) | 5 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 4 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 22 | 7 | 0
Neutropenia (Blood and lymphatic system disorders) | 6 | 2 | 0
Vision blurred (Eye disorders) | 3 | 2 | 0
Anorexia (Metabolism and nutrition disorders) | 6 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 4 | 3 | 0
Haemoglobin decreased (Investigations) | 2 | 2 | 0
Blood triglycerides increased (Investigations) | 1 | 2 | 0
Hypertension (Vascular disorders) | 0 | 3 | 0
Dry mouth (Gastrointestinal disorders) | 2 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days